CLINICAL TRIAL: NCT03139682
Title: Microvascular Injury and Blood-brain Barrier Dysfunction as Novel Biomarkers and Targets for Treatment in Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Other Study IDs: TMI_BBBD_2017
Record Dates: First submitted 2017-04-26; First posted 2017-05-04 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Traumatic Brain Injury; Blood Brain Barrier Defect
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum tau protein (sTau), von Willebrand factor (vWF), brain derived neurotrophic factor (BDNF), glial fibrillary acidic protein (GFAP),S100β, and serum neurofilament light (sNFL).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death and disability around the world. The social and economic burden of TBI is tremendous and the cost of TBI is estimated at $1 billion per year in Canada- $650 million in care and $580 million in lost productivity. Novel interventions aimed at TBI-linked molecular targets have been successful in limiting injury and improving neurologic recovery in animal models, thus providing compelling evidence that effective intervention is possible after injury. This study proposes to investigate traumatic microvascular injury (TMI) and specifically blood-brain barrier dysfunction (BBBD) as a candidate biomarker and therapeutic target in TBI.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 85 inclusive
* Clinically diagnosed TBI or evidence of TBI
* For mild TBI, as defined by the American Congress on Rehabilitation Medicine (1993), clear evidence and/or documentation of blunt head injury and any one of the following:

  * any loss of consciousness up to 30 min
  * any loss of memory for events immediately before or after the injury as much as 24 h
  * any alteration of mental state at the time of the injury
  * focal neurologic deficits that might or might not be transient

but where the severity of the injury does not exceed oss of consciousness exceeding 30 min, posttraumatic amnesia longer than 24 h, a Glasgow Coma Scale score falling below 13 after 30 min.

* For moderate TBI (GCS 9-12) and severe TBI (GCS 4-8) CT evidence of TBI-linked abnormality (intracranial lesion including traumatic SAH, contusion, extra-axial hematoma). For patients who are intubated, use best documented GCS within first 48 hours of injury.
* Stable respiratory or hemodynamic status allowing MRI within 2-4 days of TBI as determined by the attending physician
* Patient or substitute decision maker can provide consent

Exclusion Criteria:

* Pre-existing known neurologic, psychiatric disease (dementia, prior severe TBI, schizophrenia, uncontrolled epilepsy, major depressive disorder, stroke, multiple sclerosis, brain tumor)
* Serious infection, complications (sepsis, multilobe pneumonia, etc.) < 4 days after TBI
* Acute ischemic heart disease (MI or unstable angina)
* SBP < 100 mm Hg, DBP < 60 mm Hg
* MRI contraindications; patient has metal implant, pacemaker, biostimulator, neurostimulator, internal defibrillator, history of metal in eye, inner ear implant, cerebral aneurism clip, joint replacement, any known metal in their body, or are pregnant or breast feeding
* History or evidence of active malignancy
* History or evidence of serious kidney (GFR =<60) , heart, or liver disease
* Pregnant or breast-feeding women
* Inability to complete follow up visits (e.g. tourists)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit mild (n=40), moderate (n=40) and severe (n=40) TBI patients with a TBI-linked abnormality (e.g. epidural & subdural hematomas, subarachnoid hemorrhage, contusions). TBI will be classified by severity using the Glasgow Coma Scale (GCS); mild TBI (GCS13-15), moderate TBI (GCS 9-12), and severe TBI (GCS <8).
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Change in brain volume with blood brain barrier dysfunction | At < 4, 10 ± 2, and 90 ± 10 days post-injury
  Measurement of change in brain volume with BBBD and extent of permeability change as measured by DCE-MRI
Change in serum biomarkers of blood brain barrier dysfunction | At < 4, 10 ± 2, and 90 ± 10 days post-injury
  Measurement of change in serum biomarkers of BBBD / neural injury (vWF, BDNF, GFAP, S100β, sTau, and sNFL)
Change in Glasgow Outcome Scale-Extended (GOS-E) | At 10 ± 2 days, 90 ± 10 days, and 1 year post-injury
  The GOS-E is intended to provide a general index of overall outcome that is sensitive to small but clinically relevant treatment effects in people who sustain TBI.
Change in Rivermead Post Concussion Symptom Questionnaire (RPSQ) | At 10 ± 2 days, 90 ± 10 days, and 1 year post-injury
  The RPSQ is a 16-item self-report measure administered to individual(s) who sustained a TBI in order to measure the severity of symptoms and assess progress.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) | At 10 ± 2 days, 90 ± 10 days, and 1 year post-injury
  PROMIS is a set of person-centered measures that evaluates and monitors domains such as physical, mental and social health in adults and children. For this study, we will utilize the following domains: depression, fatigue, and pain interference.
Change in post-traumatic epilepsy | At 10 ± 2 days, 90 ± 10 days, 1 year, and 2 years post-injury
  Screening for post-traumatic epilepsy

CONTACTS AND LOCATIONS:
Overall Officials: David B. Clarke, MD, PhD, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada